CLINICAL TRIAL: NCT03015909
Title: A Multi-center, Open, Single-arm, Switch-over, Prospective, Phase IV Study to Assess the Ease of Use, Preference, and Safety After 8 Weeks Subcutaneous Administration of EutropinPen Inj. in Patients Pretreated With Recombinant Human Growth Hormone by Reusable Device
Brief Title: Evaluation of the Ease of Use, Preference, and Safety of EutropinPen Inj.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LG-HGCL008
Record Dates: First submitted 2016-11-10; First posted 2017-01-10 (Estimated); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Short Stature, Idiopathic; Infant, Small for Gestational Age; Growth Hormone Deficiency; Chronic Renal Failure; Turner Syndrome
MeSH Terms: conditions — Dwarfism; Dwarfism, Pituitary; Kidney Failure, Chronic; Turner Syndrome | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eutropin pen inj. (Other)
  Interventions: Drug: Somatropin

INTERVENTIONS:
Drug: Somatropin

SUMMARY:
The purpose of this study is to assess the ease of use, preference, and safety after 8 weeks subcutaneous administration of EutropinPen Inj. in patients pretreated with recombinant human growth hormone by reusable device.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who has been using reusable device growth hormone injection in recent 3 months at least for 6 weeks
* Subjects who meets the indication of EutropinPen inj.

Exclusion Criteria:

* Subjects who has diseases below on screening visit

  * Diabetes
  * Malignant tumor
  * Epiphyseal closure
  * Chronic kidney disease (recieved kidney transplantation)
  * Acute respitory failure

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 116 (Actual)
Dates: Start 2016-08-11 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
Ease of use for EutropinPen Inj. against previous reusable device assessed by a questionnaire. | Day 57
Preference for EutropinPen Inj. against previous reusable device assessed by a questionnaire. | Day 57

SECONDARY OUTCOMES:
Benefits of EutropinPen inj. assessed by a questionnaire | Day 57
  1. Ease of use
  2. Unit
  3. High dose packing
  4. Grip
  5. Design
  6. Less pain
Fear assessed by a questionnaire | Screening, Day 57
  Ask of fearness how the child feels about the needle
Ease of use for EutropinPen Inj. at each injection step assessed by a questionnaire | Screening, Day 57
  1. Ask ease of use at each injection step (1~5 pts)
  2. Preparation time for injection
Treatment compliance of EutropinPen Inj. (%) | Day 57

CONTACTS AND LOCATIONS:
Locations (1):
- Ajou university hospital, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee JE, Kim SY, Yoo JH, Hwang IT, Lim JS, Yi KH, Rhie YJ, Lee GM, Nam HK, Chae HW, Kim EY, Cheon CK, Lee J, Shim YS, Lee Y, Kim EY, Hwang JS. Ease of Use, Preference, and Safety of the Recombinant Human Growth Hormone Disposable Pen Compared with the Reusable Device: A Multicenter, Single-Arm, Open-Label, Switch-Over, Prospective, Phase IV Trial. Patient Prefer Adherence. 2019 Dec 20;13:2195-2205. doi: 10.2147/PPA.S229536. eCollection 2019. PMID 31908426